CLINICAL TRIAL: NCT05001984
Title: Trial of PCSK9 Inhibition in Patients with Acute Stroke and Symptomatic Intracranial Atherosclerosis - a Prospective, Randomized, Open-label, Blinded End-point Study with High-resolution MR Vessel Wall Imaging
Brief Title: Trial of PCSK9 Inhibition in Patients with Acute Stroke and Symptomatic Intracranial Atherosclerosis
Acronym: TOPICAL-MRI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOPICAL-MRI; MOST 110-2314-B-182A-072 (Other Grant/Funding Number: Ministry of Science and Technology, Taiwan)
Record Dates: First submitted 2021-07-22; First posted 2021-08-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Intracranial Atherosclerosis; Acute Ischemic Stroke; ICAS - Intracranial Atherosclerosis
Keywords: Intracranial Atherosclerosis; Acute Ischemic Stroke; PCSK9 inhibitor
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemic Stroke | interventions — alirocumab

STUDY DESIGN:
Intervention Model Description: randomized, open-label, blinded end-point study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Active Comparator): In addition to high-intensity statin and antiplatelet treatment, patients will receive treatment of alirocumab 75mg subcutaneously every 2 weeks for a total of 26 weeks
  Interventions: Drug: Alirocumab
- Control group (No Intervention): Patient will have high-intensity statin and antiplatelet treatment.

INTERVENTIONS:
Drug: Alirocumab — Alirocumab 75mg subcutaneously every 2 weeks for a total of 26 weeks.
  Other Names: Praluent
  Arms: Intervention group

SUMMARY:
This study will evaluate whether low-density lipoprotein (LDL-C) lowering with alirocumab results in greater change from baseline in intracranial atherosclerotic plaque at week 26 than control in adults with acute ischemic stroke from intracranial atherosclerosis taking lipid lowering therapy.

DETAILED DESCRIPTION:
In this trial, we will conduct a prospective, randomized, open-label, blinded end-point study using high-resolution MRI in patients with acute ischemic stroke from intracranial atherosclerosis to evaluate the efficacy and safety of alirocumab. We hypothesis that additional alirocumab treatment on a background of statin therapy could result in greater stabilization of intracranial plaque and regression of arterial stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic stroke with National Institutes of Health Stroke Scale (NIHSS) score of 1-15
* Ischemic lesions on diffuse-weighted imaging located in the territory of symptomatic intracranial atherosclerosis (ICAS).
* Symptomatic ICAS (above 30%) at the M1 or M2 of the middle cerebral artery, basilar artery or at the intracranial portion of the internal carotid artery or vertebral artery.
* Serum LDL-C ≥70 mg/dL for subjects on lipid-lowering therapies (such as a statin and/or ezetimibe) or LDL-C ≥100 mg/dL for subjects without lipid-lowering therapies.
* Ability to randomize within 7 days of time last known free of new ischemic symptoms.
* Ability to receive alirocumab or statin treatment within 7 days of stroke onset.
* Head CT or MRI ruling out hemorrhage or other pathology, such as vascular malformation, tumor, or abscess, that could explain symptoms or contraindicate therapy.
* Pre-stroke modified Rankin Scale (mRS)≦2

Exclusion Criteria:

* Age <20 years.
* Judged by clinical physician.
* After endovascular intervention or endarterectomy for the symptomatic ICAS.
* Patients with more than 50% stenosis of extra-cranial arteries the relevant arteries on magnetic resonance angiography (MRA), including extra-cranial carotid artery or vertebral arteries.
* Patients with high risk of cardioembolic source, such as atrial fibrillation, acute myocardial infarction, severe heart failure or valvular heart disease.
* Other determined stroke etiology, such as vasculitis, shock, antiphospholipid antibody syndrome, arterial dissection, CADASIL and etc.
* Qualifying ischemic event induced by angiography or surgery.
* Severe non-cardiovascular comorbidity with life expectancy <6 months.
* Contraindication or allergy to alirocumab or Gadolinium
* Severe renal (serum creatinine >2 mg/dL) or calculated glomerular filtration rate <30 mL/min/ 1.73 m2 by estimated glomerular filtration rate (eGFR) using Cockcroft Gault methodology.
* Hepatic insufficiency (INR>1.2; ALT>40 U/L or any resultant complication, such as variceal bleeding, encephalopathy, or jaundice)
* Hemostatic disorder or systemic bleeding in the past 3 months
* Current thrombocytopenia (platelet count <100 x109/L) or leukopenia (<2 x109/L)
* Anemia（<10 mg/dL）
* History of drug-induced hematologic or hepatic abnormalities
* History of malignancy that required surgery, radiation therapy or systemic therapy.
* Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use effective contraception.
* Other neurological conditions that would complicate assessment of outcomes during follow-up.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
The changes of intracranial atherosclerotic plaque: stenosis degree | 26 weeks
  The changes of intracranial atherosclerotic plaque in vessel-wall MRI before and after 6-month treatment, measured as stenosis degree.
  The degree of stenosis was calculated as: (1-lumen area of stenotic lesion/reference lumen area)×100%.
The changes of intracranial atherosclerotic plaque: percent atheroma volume | 26 weeks
  The changes of intracranial atherosclerotic plaque in vessel-wall MRI before and after 6-month treatment, measured as percent atheroma volume (PAV).
  The PAV was calculated using the following equation:
  PAV = Σ(EEM area - Lumen area) / ΣEEM area × 100, where EEM area is the cross-sectional area of the external elastic membrane and Lumen area is the cross-sectional area of the lumen.
The changes of intracranial atherosclerotic plaque: enhancement volume | 26 weeks
  The changes of intracranial atherosclerotic plaque in vessel-wall MRI before and after 6-month treatment, measured as enhancement volume.
  The enhancement volume was measured as post-contrast plaque enhancement for intracranial arteries and intraplaque hemorrhage.

SECONDARY OUTCOMES:
Percentage of patients with major cardiovascular events | 26 weeks
  Defined as the composite of cardiovascular death, myocardial infarction, transient ischemic attack, ischemic stroke and hemorrhagic stroke.
Percentage of patients with myocardial infarction | 26 weeks
  patients with myocardial infarction
Percentage of patients with cardiovascular death | 26 weeks
  patients with cardiovascular death
Percentage of patients with stroke | 26 weeks
  Include transient ischemic attack, ischemic and hemorrhagic stroke
Percentage of patients with ischemic stroke or transient ischemic attack. | 26 weeks
  Percentage of patients with ischemic stroke or transient ischemic attack.
Percentage of patients with new ischemic lesions | 26 weeks
  Defined as new ischemic lesions in the territory of ICAS between 2 MRIs
Percentage of patients with favorable functional recovery | 3 months
  Defined as a mRS ≦2 mRS. The Modified Rankin Scale (mRS) runs from 0-6, running from perfect health without symptoms(score 0) to death(score 6).
Changes in serum biomarkers | 26 weeks
  Include liver function tests, HbA1c and lipid profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Yenchu Huang, MD, Study Director — Chang Gung Memorial Hospital, Chiayi
Locations (1):
- Yenchu Huang, Chiayi City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmstedt CA, Turan TN, Chimowitz MI. Atherosclerotic intracranial arterial stenosis: risk factors, diagnosis, and treatment. Lancet Neurol. 2013 Nov;12(11):1106-14. doi: 10.1016/S1474-4422(13)70195-9. PMID 24135208
- [Background] Wang Y, Zhao X, Liu L, Soo YO, Pu Y, Pan Y, Wang Y, Zou X, Leung TW, Cai Y, Bai Q, Wu Y, Wang C, Pan X, Luo B, Wong KS; CICAS Study Group. Prevalence and outcomes of symptomatic intracranial large artery stenoses and occlusions in China: the Chinese Intracranial Atherosclerosis (CICAS) Study. Stroke. 2014 Mar;45(3):663-9. doi: 10.1161/STROKEAHA.113.003508. Epub 2014 Jan 30. PMID 24481975
- [Background] Hurford R, Wolters FJ, Li L, Lau KK, Kuker W, Rothwell PM; Oxford Vascular Study Phenotyped Cohort. Prevalence, predictors, and prognosis of symptomatic intracranial stenosis in patients with transient ischaemic attack or minor stroke: a population-based cohort study. Lancet Neurol. 2020 May;19(5):413-421. doi: 10.1016/S1474-4422(20)30079-X. PMID 32333899
- [Background] Gao S, Wang YJ, Xu AD, Li YS, Wang DZ. Chinese ischemic stroke subclassification. Front Neurol. 2011 Feb 15;2:6. doi: 10.3389/fneur.2011.00006. eCollection 2011. PMID 21427797
- [Background] Xu W. High-resolution MRI of intracranial large artery diseases: how to use it in clinical practice? Stroke Vasc Neurol. 2019 Jun 20;4(2):102-104. doi: 10.1136/svn-2018-000210. eCollection 2019 Jul. PMID 31338221
- [Background] Xu WH, Li ML, Gao S, Ni J, Yao M, Zhou LX, Peng B, Feng F, Jin ZY, Cui LY. Middle cerebral artery intraplaque hemorrhage: prevalence and clinical relevance. Ann Neurol. 2012 Feb;71(2):195-8. doi: 10.1002/ana.22626. PMID 22367991
- [Background] Petrone L, Nannoni S, Del Bene A, Palumbo V, Inzitari D. Branch Atheromatous Disease: A Clinically Meaningful, Yet Unproven Concept. Cerebrovasc Dis. 2016;41(1-2):87-95. doi: 10.1159/000442577. Epub 2015 Dec 16. PMID 26671513
- [Background] Yamamoto Y, Ohara T, Hamanaka M, Hosomi A, Tamura A, Akiguchi I. Characteristics of intracranial branch atheromatous disease and its association with progressive motor deficits. J Neurol Sci. 2011 May 15;304(1-2):78-82. doi: 10.1016/j.jns.2011.02.006. Epub 2011 Mar 13. PMID 21402390
- [Background] Kim JS, Yoon Y. Single subcortical infarction associated with parental arterial disease: important yet neglected sub-type of atherothrombotic stroke. Int J Stroke. 2013 Apr;8(3):197-203. doi: 10.1111/j.1747-4949.2012.00816.x. Epub 2012 May 9. PMID 22568537
- [Background] Liu D, Liu J, Cai Y, Wong KSL, Liu L. Is the future of symptomatic intracranial atherosclerotic stenosis management promising? J Neurol Neurosurg Psychiatry. 2020 Feb;91(2):122-124. doi: 10.1136/jnnp-2019-321564. No abstract available. PMID 31919104
- [Background] Johnston SC, Easton JD, Farrant M, Barsan W, Conwit RA, Elm JJ, Kim AS, Lindblad AS, Palesch YY; Clinical Research Collaboration, Neurological Emergencies Treatment Trials Network, and the POINT Investigators. Clopidogrel and Aspirin in Acute Ischemic Stroke and High-Risk TIA. N Engl J Med. 2018 Jul 19;379(3):215-225. doi: 10.1056/NEJMoa1800410. Epub 2018 May 16. PMID 29766750
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Background] Kim D, Park JM, Kang K, Cho YJ, Hong KS, Lee KB, Park TH, Lee SJ, Kim JG, Han MK, Kim BJ, Lee J, Cha JK, Kim DH, Nah HW, Kim DE, Ryu WS, Kim JT, Choi KH, Choi JC, Lee BC, Yu KH, Oh MS, Kim WJ, Kwon JH, Shin DI, Sohn SI, Hong JH, Lee JS, Lee J, Gorelick PB, Bae HJ. Dual Versus Mono Antiplatelet Therapy in Large Atherosclerotic Stroke. Stroke. 2019 May;50(5):1184-1192. doi: 10.1161/STROKEAHA.119.024786. PMID 30932785
- [Background] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Background] Weinberger J. Comparison of warfarin and aspirin for symptomatic intracranial arterial stenosis. Curr Cardiol Rep. 2006 Feb;8(1):7. No abstract available. PMID 16507227
- [Background] Amarenco P, Bogousslavsky J, Callahan A 3rd, Goldstein LB, Hennerici M, Rudolph AE, Sillesen H, Simunovic L, Szarek M, Welch KM, Zivin JA; Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) Investigators. High-dose atorvastatin after stroke or transient ischemic attack. N Engl J Med. 2006 Aug 10;355(6):549-59. doi: 10.1056/NEJMoa061894. PMID 16899775
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] Schwartz GG, Steg PG, Szarek M, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Pordy R, Quintero K, Roe MT, Sasiela WJ, Tamby JF, Tricoci P, White HD, Zeiher AM; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab and Cardiovascular Outcomes after Acute Coronary Syndrome. N Engl J Med. 2018 Nov 29;379(22):2097-2107. doi: 10.1056/NEJMoa1801174. Epub 2018 Nov 7. PMID 30403574
- [Background] Hadjiphilippou S, Ray KK. Evolocumab and clinical outcomes in patients with cardiovascular disease. J R Coll Physicians Edinb. 2017 Jun;47(2):153-155. doi: 10.4997/JRCPE.2017.212. No abstract available. PMID 28675189
- [Background] Huynh K. Dyslipidaemia. Assessing the efficacy and safety of evolocumab and alirocumab. Nat Rev Cardiol. 2015 May;12(5):261. doi: 10.1038/nrcardio.2015.51. Epub 2015 Mar 31. No abstract available. PMID 25824512
- [Background] Chung JW, Cha J, Lee MJ, Yu IW, Park MS, Seo WK, Kim ST, Bang OY. Intensive Statin Treatment in Acute Ischaemic Stroke Patients with Intracranial Atherosclerosis: a High-Resolution Magnetic Resonance Imaging study (STAMINA-MRI Study). J Neurol Neurosurg Psychiatry. 2020 Feb;91(2):204-211. doi: 10.1136/jnnp-2019-320893. Epub 2019 Aug 1. PMID 31371644
- [Derived] Huang YC, Chang CH, Tsai YH, Weng HH, Lin LC, Lee JD. PCSK9 inhibition in patients with acute stroke and symptomatic intracranial atherosclerosis: protocol for a prospective, randomised, open-label, blinded end-point trial with vessel-wall MR imaging. BMJ Open. 2022 Apr 29;12(4):e060068. doi: 10.1136/bmjopen-2021-060068. PMID 35487727